CLINICAL TRIAL: NCT06887595
Title: A Comparative Study of AI-Powered/Computer-Guided Versus Conventional Linear Micro-Perforation Split Approach for Treatment of Horizontal Mandibular Ridge Atrophy (A Randomized Clinical Trial)
Brief Title: Linear Micro-Perforation Ridge Split Approach
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Walid Elamrousy, Assistant Professor of periodontology, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KFSIRB200-467
Record Dates: First submitted 2025-03-16; First posted 2025-03-20 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Alveolar Bone Loss; Dental Implant Failed
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group I (Experimental): ridge split and expansion with free-hand linear micro perforation osteotomy approach with simultaneous implant placement
  Interventions: Procedure: Free-hand linear micro perforation osteotomy and ridge splitting
- study group II (Experimental): ridge split and expansion with AI-assisted/computer-guided (linear micro perforation osteotomy approach with simultaneous implant placement)
  Interventions: Procedure: AI-assisted/computer-guided linear micro perforation osteotomy and ridge splitting

INTERVENTIONS:
Procedure: Free-hand linear micro perforation osteotomy and ridge splitting — AI-assisted/computer-guided linear micro perforation osteotomy and ridge splitting
  Other Names: Free-hand crestal ridge splitting expansion after linear micro perforation osteotomy will be performed using electromagnetic mallet
  Arms: study group I
Procedure: AI-assisted/computer-guided linear micro perforation osteotomy and ridge splitting — AI-assisted/computer-guided crestal ridge splitting expansion after linear micro perforation osteotomy will be performed using electromagnetic mallet
  Arms: study group II

SUMMARY:
The traditional ridge split technique might be performed simultaneously with implant placement, resulting in a shortened treatment time. However, this approach has the potential for serious complications, including buccal bone fracture, prolonged pain or paresthesia, and loss of bone height. Linear Micro-Perforation Osteotomy (LMPO) has emerged as a less invasive alternative, promoting natural bone expansion through controlled micro-perforations in the cortical bone, allowing for ridge widening without extensive grafting. However, the precision required for LMPO can be difficult to achieve manually, especially in anatomically complex or narrow ridge areas, leading to variability in outcomes and potential risks such as bone fractures or inadequate expansion.Our study aims to evaluate the efficacy, clinical, and radiological outcomes of the flapless AI-powered/computer-guided LMPO ridge split/expansion technique compared to the traditional LMPO ridge split/expansion method for lateral ridge reconstruction of mandibular horizontal ridge deficiencies.

DETAILED DESCRIPTION:
In contemporary dentistry, the aim is to replace missing teeth with prosthetics or to remove diseased teeth from the patient and return them to normal in terms of shape, function, comfort, appearance, speech, and health. Why implant dentistry is different is the capacity to fulfill this objective despite atrophy, illness, or harm to the stomatognathic apparatus.

Implant-based dental rehabilitation of partly or completely edentulous areas has become a frequent procedure with consistent long-term outcomes in recent decades. Nevertheless, alveolar ridges are frequently impaired with horizontal inadequacy as a result of bone resorption, which has an impact on implant application.

The resorption of alveolar bone is a common sequelae of tooth loss and presents a clinical problem for implant placement. Implants must be placed with at least 1 mm of bone on the buccal and lingual aspects to maintain crestal bone levels.

Narrow edentulous ridges less than 5 mm wide present a challenge to the clinician for implant placement. Hence, lateral bone augmentation procedures are necessary to overcome maxillary and mandibular bone deficiencies. These procedures involve the use of bone augmentation, such as guided bone regeneration (GBR), bone block (autogenous or non-autogenous), and conventional onlay/inlay graft. Those procedures have many drawbacks such as longer healing time (6-9 months) for adequate bone regeneration before implant placement, the possibility of membrane exposure, an increased risk of infection, high cost, and rapid graft resorption; thus leading to inadequate bone regeneration or loss of the newly formed bone.

Based on previous knowledge, ridge split/expansion was introduced as an alternative to treat the width insufficiency of alveolar ridges with specific indications. The basic procedure includes a sagittal osteotomy in the center of the edentulous ridge, where the two cortical plates are expanded to increase the width and thereby simultaneous implant insertion with an appropriate diameter could be achieved.

Due to double cellularity and double vascularity gained from the lateral bony plate, bone healing, and regeneration tendency were significantly improved without the need for bone graft or membrane. A shorter treatment period, no need for donor sites, and the possibility of simultaneous implant placement are among the merits of ridge splitting over different augmentation techniques.

For successful ridge split with simultaneous implantation, the alveolar ridge width should be 3 mm or more with at least 1 mm trabecular bone between the cortical plates.

The splitting could be performed using the chisel and mallet, the surgical disc, ultra-fine fissure burs, and recently the piezoelectric surgical devices and the electromagnetic mallet. Osteotomes, chisels, bone spreaders, and engine-driven expanders were utilized for Ridge expansion.

The traditional ridge split technique might be performed simultaneously with implant placement, resulting in a shortened treatment time. However, this approach has the potential for serious complications, including buccal bone fracture, prolonged pain or paresthesia, and loss of bone height. On the other hand, the staged approach has been proposed with splitting and expansion performed followed by implant placement after a 3-week healing interval to allow re-establishment of the blood supply to the surgical site.

Linear Micro-Perforation Osteotomy (LMPO) has emerged as a less invasive alternative, promoting natural bone expansion through controlled micro-perforations in the cortical bone, allowing for ridge widening without extensive grafting. However, the precision required for LMPO can be difficult to achieve manually, especially in anatomically complex or narrow ridge areas, leading to variability in outcomes and potential risks such as bone fractures or inadequate expansion.

Computer-guided technology presents an opportunity to enhance LMPO by providing a structured, pre-planned guide for split-osteotomy and expansion. Utilizing 3D imaging data, a computer-guided splint can be custom-fabricated to fit each patient's unique anatomy, offering unparalleled accuracy in osteotomy execution and minimizing the risk of error. Additionally, performing LMPO without flap elevation with the assistance of this guided splint further reduces surgical trauma, preserves periosteal blood supply, and promotes faster healing, making it a more patient-friendly option.

Limited clinical data are available about LMPO. Our study aims to evaluate the efficacy, clinical, and radiological outcomes of the flapless AI-powered/computer-guided LMPO ridge split/expansion technique compared to the traditional LMPO ridge split/expansion method for lateral ridge reconstruction of mandibular horizontal ridge deficiencies.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with narrow alveolar ridge that requires dental implantation.

  * Minimum bone width of 3 mm
  * Ridge width of not less than 3 mm in CBCT image
  * Minimum bone height of 10 mm
  * Proper inter-occlusal space
  * Perioperative cone beam CT scan image of the atrophic ridge

Exclusion Criteria:

* • Uncontrolled diabetes.

  * Heavy smokers.
  * Current chemotherapy or radiotherapy.
  * Alcohol or drug abuse.
  * Pregnant women.
  * Active infection.
  * Inter-occlusal space not less than 7-8 mm.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2025-03-18 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
ridge width | 12-months
  The width of the alveolar bone will be measured again using CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry, kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided